CLINICAL TRIAL: NCT01753622
Title: Effect of a Supervised Exercise Program in Obese and Overweight Pregnant Women on Outcomes and Level of Depression. A Randomized Controlled Trial
Brief Title: Physical Exercise Program in Obese and Overweight Pregnant Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technical University of Madrid (Other)
Responsible Party: Principal Investigator, María Perales Santaella, PhD student, Technical University of Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Overweight-obese pregnant
Record Dates: First submitted 2012-12-17; First posted 2012-12-20 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2012-12

CONDITIONS: Pregnancy
Keywords: Overweight, obese, pregnant, depression, outcomes
MeSH Terms: conditions — Overweight; Obesity; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention): Sedentary Obese and overweight pregnant women
- Exercise group (Experimental): Physical exercise program
  Interventions: Behavioral: Exercise group

INTERVENTIONS:
Behavioral: Exercise group — Supervised physical conditioning program of three 55-60 minute sessions per week during whole pregnancy (from week 9 to 38). Each session consists of 25-30 minutes of cardiovascular exercise, 10 minutes of specific exercises (strength and balance exercises), and 10 minutes of pelvic floor muscles training.
  Aerobic activity was prescribed at light to moderate intensity, aiming for 55-60 of maximal heart rate. All subjects wore a heart rate (HR) monitor (Polar FT7) during the training sessions to ensure that exercise intensity was light to moderate.
  Arms: Exercise group

SUMMARY:
Obesity and overweight have become an epidemic in the world and its prevalence between pregnant women is especially dangerous. Having a high Body Mass Index (BMI) is also associated with depression disorders and its serious complications during this period.

DETAILED DESCRIPTION:
The aim of our study is to assess whether a specific exercise program during pregnancy has a positive effect on maternal mood and other pregnancy outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Being healthy and able to exercise following American College of Obstetricians and Gynecologists (ACOG) guidelines
* Being able to communicate in spanish
* Giving birth at Hospital Universitario de Fuenlabrada
* Having a Body Mass Index (BMI) greater than 24.9

Exclusion Criteria:

* Multiparity
* Obstetrician complications
* Being interested in the study after 18 weeks
* Not being regular in physical exercise program (minimum adherence 80%)
* Younger than 18 years old

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2009-10; Primary Completion 2013-01 (Actual); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Change from level of depression at the end of the pregnancy | Up to 36 weeks
  The Center for Epidemiological Studies-Depression scale (CES-D) was administered to all obese and overweight pregnant women at the beginning and at the end of their pregnancies

SECONDARY OUTCOMES:
Maternal gestational weight gain | 40-42 weeks
  Maternal gain weight
Maternal outcomes | After labor
  Type of labor

OTHER OUTCOMES:
Fetal weight | After labor
  Birth weight (g.)

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Barakat, PhD, Study Director — Universidad Politecnica de Madrid
Locations (1):
- Universidad Politecnica de Madrid, Madrid, Madrid, Spain